CLINICAL TRIAL: NCT06394310
Title: The Effectiveness of Dry Needling on Reducing Spasticity and Promoting Mobility and Balance in People With Multiple Sclerosis
Brief Title: Dry Needling in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jacob J. Sosnoff, Ph.D., Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00151015
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Spasticity
Keywords: multiple sclerosis; Dry needling; Spasticity; Mobility; Balance
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry needling (Experimental): Participants will complete three sessions of dry needling through three weeks (one session per each week)
  Interventions: Device: Dry needling
- Sham DN (Sham Comparator): Participants randomized to the control group will be receiving sham needling
  Interventions: Device: Sham dry needling

INTERVENTIONS:
Device: Dry needling — The dry needling technique will employ in the current proposed study follows the standard technique for needling patients with spasticity
  Arms: Dry needling
Device: Sham dry needling — In the control group, The investigators will use the methods proposed by Cushman et al. to apply sham dry needling (DN) to our participants
  Arms: Sham DN

SUMMARY:
The investigators are doing this study to see if a treatment called dry needling improves muscle spasticity (muscle tightness) in people who have Multiple Sclerosis. Dry needling involves using tiny needles, like those in acupuncture, to target some muscles, like calf muscles. It differs from traditional acupuncture as it focuses on treating or managing muscle spots, aiming to reduce muscle stiffness and pain. Dry needling may offer a minimally-invasive and medication-free approach to improve muscle spasticity. The investigators hope to see if dry needling also helps enhance balance and walking abilities. This might provide potential improvements inoverall mobility and balance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 64 years
* Clinical diagnosis of Multiple Sclerosis based on the McDonald Criteria
* Spasticity in their lower legs
* Patient Determined Disease Steps (PDDS) score of 5 or below

Exclusion Criteria:

* Inability to communicate effectively with study personnel
* Needle phobia
* Severe varicose veins
* Presence of an active implanted device
* Pregnancy
* Any active cancer or history within 1 year
* known or suspected infection at the site of needling or in the surrounding area
* Presence of a fixed plantarflexion contracture at the ankle
* Acute fracture of dislocation in the region (bilateral lower extremity)
* Deep vein thrombosis or peripheral vascular disease
* Thrombophlebitis, or active osteomyelitis in the region (bilateral lower extremity)
* Any medication changes, including antispastic medicines, for the past three months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-02 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Spasticity | 5 weeks
  Spasticity will be assessed through the Modified Ashworth scale (Scored between 0 to 4, with higher scores show higher level of spasticity)

CONTACTS AND LOCATIONS:
Locations (1):
- Mobility and Falls Lab, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided